CLINICAL TRIAL: NCT02529085
Title: Study of Early Endocrine Profile in Infants With Prader-Willi Syndrome (PWS) in Order to Unravel the Switch From Early Feeding Difficulties to Obesity and Hyperphagia.
Brief Title: PWS European Blood Bank for Infants and Controls From 0 to 48 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: European Society for Paediatric Endocrinology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12 359 03
Record Dates: First submitted 2015-04-24; First posted 2015-08-19 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infants with PWS (Experimental): Blood samples for the bank in link with a multicenter database including clinical data on birth, auxology, endocrine functions and feeding behaviour
  Interventions: Other: blood samples
- control group (Other): Blood samples for the bank in children hospitalized for a planned surgery for malformation, orthopaedic or visceral surgery
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — blood samples for the bank

SUMMARY:
The present project aims to determine the underlying mechanisms for the switch from failure to thrive to excessive weight gain and hyperphagia with impaired satiety in PWS. The primary objective is to describe the evolution of circulating hormones involved in feeding and appetite regulation during the 4 first years of life. The secondary objective is to make this blood bank available for other research projects and particularly the investigation of hormones involved in hypogonadism.

Over the last ten years, the age at diagnosis in PWS has fallen significantly and the majority of cases is now diagnosed during the 1st trimester of life giving the possibility to collect precise clinical data and serum samples at early stages. The investigators of the project are involved in the care of patients with PWS and have a devoted clinic and an organized network in their country through clinical networks or patient associations.

DETAILED DESCRIPTION:
The investigators propose to perform a prospective multicentric study, both longitudinal (duration 30 months) and cross-sectional with implementation of a blood bank in link with a multicenter database including clinical data on birth, auxology, endocrine functions and feeding behaviour. The cohort will include 200 infants from 3 to 48 months with PWS and 200 controls matched on age recruited in the 6 participating countries. The investigators make the assumption that 3 blood sampling will be necessary during the first year and 6 monthly sampling thereafter. For measuring hormones and neuropeptides (ghrelin, insulin, leptin, pancreatic polypeptide, oxytocin, cortisol, melatonin, orexin A, GLP-1 and PYY) involved in feeding and appetite regulation the investigators will use primarily multiplex microplates technics requiring 50-200µl of sample. Intragroup and intergroup comparisons will be performed in order to describe the evolution of each hormone with time and to compare data obtained in the PWS group with those obtained in the control group.

ELIGIBILITY:
Inclusion Criteria (PWS infants cohort)

* Genetic diagnosis of Prader-Willi syndrome

Exclusion Criteria (PWS infants cohort)

* none

Inclusion Criteria (control group)

* children hospitalized for a planned surgery for malformation, orthopaedic or visceral surgery

Exclusion Criteria (control group)

* children with endocrine disorder

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 215 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Levels of hormones and neuropeptides | 42 months
  Measure of hormones and neuropeptides (ghrelin, insulin, leptin, pancreatic polypeptide, oxytocin, melatonin, orexins) involved in feeding and appetite regulation

SECONDARY OUTCOMES:
Correlation between hormones and neuropeptides levels | 42 months
  study the correlation between ghrelin, insulin, leptin, pancreatic polypeptide, oxytocin, melatonin, orexins

CONTACTS AND LOCATIONS:
Overall Officials: Maithe TAUBER, MD, Principal Investigator — University Hospital, Toulouse
Locations (6):
- Unité d'Endocrinologie Pédiatrique / Université Catholique de Louvain, Brussels, Belgium
- Department of Pediatrics / Division of Endocrinology, Toulouse, Haute-Garonne, France
- Department of Endocrinology / University Children's Hospital, Essen, Germany
- Department of Pediatrics / Division of Endocrinology / Erasmus University Medical Center / Sophia Children's Hospital Rotterdam, Rotterdam, Netherlands
- Karolinska University Hospital, Stockholm, Sweden
- Metabolic & Molecular Imaging Group / MRC Clinical Sciences Centre / Imperial College London / Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Background] Cadoudal T, Buleon M, Sengenes C, Diene G, Desneulin F, Molinas C, Eddiry S, Conte-Auriol F, Daviaud D, Martin PG, Bouloumie A, Salles JP, Tauber M, Valet P. Impairment of adipose tissue in Prader-Willi syndrome rescued by growth hormone treatment. Int J Obes (Lond). 2014 Sep;38(9):1234-40. doi: 10.1038/ijo.2014.3. Epub 2014 Jan 10. PMID 24406482
- [Derived] Beauloye V, Diene G, Kuppens R, Zech F, Winandy C, Molinas C, Faye S, Kieffer I, Beckers D, Nergardh R, Hauffa B, Derycke C, Delhanty P, Hokken-Koelega A, Tauber M. High unacylated ghrelin levels support the concept of anorexia in infants with prader-willi syndrome. Orphanet J Rare Dis. 2016 May 4;11(1):56. doi: 10.1186/s13023-016-0440-0. PMID 27146407